CLINICAL TRIAL: NCT07097714
Title: Evaluating the Clinical Efficacy of Collagen Scaffold (Ossix VOLUMAX) With Piezo-Surgical Decortication in Enhancing Orthodontic Treatment Outcomes: A Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NMSI DENTMASTER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ДМ003
Record Dates: First submitted 2024-04-10; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Dental Crowding; Gingival Recession; Thin Phenotype
Keywords: Corticotomy, Soft Tissue Augmantation, Bone Augmentation, Ossix Volume, Collagene Scaffold, Orthodontics, Piezocision
MeSH Terms: conditions — Crowding; Gingival Recession

STUDY DESIGN:
Intervention Model Description: Intervention Group:
  Participants in this arm will undergo piezocisions, a minimally invasive surgical technique that aids in orthodontic tooth movement by creating vertical corticotomy grooves in the alveolar bone to facilitate its remodeling. Along with this procedure, a Collagen Scaffold will be applied. The scaffold is likely designed to support the regeneration of bone and soft tissue, potentially enhancing the effects of the decortication .
  The control group will receive piezocisions will be performed in strategic locations to accelerate as well ensuring that any effects due to the decortication process itself are not attributed to the novel treatment.Instead of the collagen scaffold, participants of this group will receive a Deepitelized Free Gingival Graft (DFGG), which is a well-established technique for increasing a soft tissue volume and treating gingival recession.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Description of Arm:
  This group will receive the novel treatment combination. Participants will undergo piezocision-a minimally invasive surgical technique that creates vertical corticotomy grooves in the alveolar bone to stimulate bone remodeling and accelerate orthodontic tooth movement. In addition, a ribose cross-linked collagen matrix (Ossix® Volumax) will be applied over the decorticated bone surface. All participants are undergoing active orthodontic treatment with fixed appliances prior to the surgical procedure.
  Intervention Name:
  Procedure/Surgery: Piezocision with ribose cross-linked collagen matrix (Ossix® Volumax)
  Intervention Description:
  A minimally invasive full-thickness flap will be elevated to expose the alveolar bone. Vertical corticotomy grooves (piezocision) will be performed in strategic locations. The collagen matrix (Ossix® Volumax) will be trimmed and applied over the exposed decorticated bone to support bone and soft tissue regeneration.
  Other Name(s):
  Interventions: Procedure: Piezocision with ribose cross-linked collagen matrix (Ossix® Volumax)
- Control (Active Comparator): Description of Arm:
  This group will receive the control treatment. Piezocision will be performed similarly to the experimental group, creating vertical corticotomy grooves to accelerate tooth movement. However, instead of a collagen matrix, participants will receive a deepithelialized free gingival graft (DFGG) harvested from the palatal mucosa. This well-established technique is commonly used to increase gingival thickness and volume and serves as a comparator for evaluating the potential added benefit of the collagen scaffold.
  Intervention Name:
  Procedure/Surgery: Piezocision with deepithelialized free gingival graft (DFGG)
  Intervention Description:
  A full-thickness mucoperiosteal flap will be elevated to expose the alveolar bone. Vertical corticotomy grooves will be created (piezocision) in strategic locations to accelerate orthodontic tooth movement. A deepithelialized free gingival graft harvested from the palate will then be placed and stabilized over the decorticated bone
  Interventions: Procedure: control

INTERVENTIONS:
Procedure: Piezocision with ribose cross-linked collagen matrix (Ossix® Volumax) — A full-thickness mucoperiosteal flap will be elevated to expose the alveolar bone. Vertical corticotomy grooves (piezocision) will be created in strategic locations to accelerate orthodontic tooth movement. The Ossix® Volumax collagen matrix will be trimmed and applied directly onto the decorticated bone surface to support bone regeneration and soft tissue augmentation.
  Other Names: Volumax; Ribose cross-linked collagen scaffold; Ossix collagen matrix
  Arms: Intervention
Procedure: control — A minimally invasive full thickness flap will be raised to expose the alveolar bone. Vertical corticotomy grooves will be performed in strategic locations to accelerate orthodontic tooth movement. The Deepitelized Free Gingival Graft (DFGG) will be placed and secured over the areas of decortication to promote soft tissue healing and augmentation.
  Arms: Control

SUMMARY:
Recent advances in orthodontic treatment have explored various materials to enhance treatment efficacy, particularly focusing on collagen scaffolds. Collagen, being a primary component of the bone matrix, has garnered attention for its biocompatibility, cell adhesion, and osteoconductivity properties. Studies have shown that collagen scaffolds undergo natural degradation, mimicking biological processes, and play a significant role in tissue engineering (International Journal of Implant Dentistry, 2023). This aligns with the growing interest in minimally invasive methods that accelerate orthodontic treatment and improve tissue regeneration.

In this context, the application of collagen scaffolds, such as Ossix VOLUMAX, in conjunction with piezo-surgical decortication, presents a novel approach. This study aims to build upon the existing knowledge, exploring the efficacy of collagen scaffolds in enhancing orthodontic treatment outcomes, especially in patients with specific dental conditions like a thin gingival phenotype and malocclusion. The study's hypothesis is grounded in the promising properties of collagen-based materials in dental and orthodontic applications, as evidenced by recent research in the field.

DETAILED DESCRIPTION:
Hypothesis:

The application of a Collagen Scaffold (Ossix VOLUMAX) in conjunction with piezo- surgical decortication enhances the efficacy of orthodontic treatment by increasing the thickness of gingiva and volume of alveolar bone in adults with a thin phenotype of gingiva and malocclusion, particularly in the mandibular incisors, more effectively than piezo- surgical decortication with a connective tissue graft alone. This combined treatment also reduces morbidity, decreases the risk of gingival recessions, and shortens the duration of surgery compared to the control group.

Study Groups:

In this clinical trial, the participants are divided into two groups to compare the outcomes of different surgical interventions in conjunction with orthodontic treatment:

Intervention Group:

This group will receive the novel treatment combination. Participants in this arm will undergo piezocisions, a minimally invasive surgical technique that aids in orthodontic tooth movement by creating vertical corticotomy grooves in the alveolar bone to facilitate its remodeling. Along with this procedure, a Collagen Scaffold (specifically, Ossix VOLUMAX) will be applied. The scaffold is likely designed to support the regeneration of bone and soft tissue, potentially enhancing the effects of the decortication and improving clinical outcomes such as bone volume and gingival thickness.

Control Group:

The control group will receive piezocisions will be performed in strategic locations to accelerate as well ensuring that any effects due to the decortication process itself are not attributed to the novel treatment.Instead of the collagen scaffold, participants of this group will receive a Deepitelized Free Gingival Graft (DFGG), which is a well-established technique for increasing a soft tissue volume and treating gingival recession. The DFGG serves as a standard comparison to evaluate the added benefit, if any of the collagen scaffold used in the intervention group.

Treatment methods:

Intervention Group: Collagen Scaffold with Piezocision

Piezcision:

Procedure: Decortication in alveolar bone was done using piezotome handpiece with piezo surgical knife, precise and selective vertical corticotomy grooves which are about 1.5-2 mm in depth will be made in the cortical bone around teeth that are targeted for movement in the interradicular area.

Technique: A minimally invasive full thickness flap will be raised to expose the alveolar bone. Vertical corticotomy grooves will be performed in strategic locations to accelerate orthodontic tooth movement.

Parameters: Vertical corticotomy grooves will be performed in strategic locations in the interradicular area which are about 1.5-2 mm in depth by gently working around the root of the tooth without damaging it, and distribution of the cuts will be standardized based on the best available evidence and will be documented for each patient.

Collagen Scaffold (Osssix VOLUMAX):

Application: After the decortication, the collagen scaffold will be applied directly onto the bone surface.

Characteristics: The scaffold is composed sugar cross-linked of byoresobable collagene 1 type (porcine), 1.5 mm thikness, resorption time 4 month.

Post-Operative Care: Standardized instructions will be provided for home care, including oral hygiene and medication, if any, to support scaffold integration.

ELIGIBILITY:
Gingival Phenotype: Participants must be diagnosed with a thin phenotype of gingiva. This could be measured using a periodontal probe to assess the thickness of the gingiva, typically less than 1 mm is considered thin. In this area may be gingival recession 1,2 Cairo type.

Dental Health: Participants must have a sufficient number of teeth and bone support to undergo orthodontic treatment. A minimum number of teeth or specific dental conditions may be outlined to ensure that the treatment can be applied effectively.

Malocclusion: Participants must be diagnosed with malocclusion, specifically requiring correction in the mandibular incisors. The type and severity of malocclusion can be classified according to a recognized system such as the Angle classification or the Index of Orthodontic Treatment Need (IOTN).

Medical History: Participants must not have any contraindications to dental surgery or orthodontic treatment, such as uncontrolled diabetes, bisphosphonate therapy, or a history of radiation to the jaws.

Consent: Participants must be able to understand the nature of the study and provide informed consent to participate in the trial.

Availability: Participants must be available for the duration of the study and able to attend all scheduled appointments for treatment and follow-up assessments.

Periodontal Health: Participants should have good periodontal health or controlled periodontitis. This may involve a preliminary periodontal assessment, ensuring that there are no active diseases that could complicate the orthodontic treatment or surgical interventions.

Orthodontic Treatment Status: Participants must not have undergone any orthodontic treatment in the past six months to ensure that any previous treatments do not affect the outcomes of the current study.

No Concurrent Dental Procedures: Participants should not be undergoing concurrent dental procedures that could affect the outcomes of the orthodontic treatment, such as implants or extensive restorative work, not coordinated with the current treatment plan Radiographic Evaluation: Suitable candidates must have clear radiographic evidence that supports the diagnosis of malocclusion and allows for the assessment of alveolar bone volume and gingival thickness. This may include recent CBCT scans or panoramic radiographs.

Non-smoker Status:

Non-smokers or individuals who have smoke less than 10 cigarettes per day may be included to avoid the confounding effects of smoking on periodontal health and healing.

Exclusion criteria:

Existing Periodontal Disease: Individuals with active periodontal disease or significant periodontal bone loss that contraindicates orthodontic treatment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2025-09-25 (Estimated); Study Completion 2026-09-25 (Estimated)

PRIMARY OUTCOMES:
Increase in Gingival Thickness and Alveolar Bone Volume | Baseline measurements will be taken prior to the surgical intervention. Subsequent measurements will be taken at 1 month, 6 months, and 1 year post-surgery. Each measurement will be conducted by blinded examiners to maintain objectivity.
  The primary endpoint is the quantifiable increase in gingival thickness and alveolar bone volume at the sites of orthodontic intervention. Gingival thickness will be defined as the distance from the gingival margin to the alveolar bone crest, and bone volume will be measured in cubic millimeters.

SECONDARY OUTCOMES:
Risk Reduction of Gingival Recession | Clinical periodontal probing and intraoral photographs will be used to measure and document changes in the gingival margin position.Measurements will be taken at baseline and at each subsequent follow-up visit, with comparison to pre-treatment levels.
  A decrease in the incidence of gingival recession post-treatment, characterized by the exposure of the roots of the teeth as measured from the cementoenamel junction (CEJ) to the gingival margin.
Decrease in Duration of Surgery | Surgical duration will be precisely recorded in minutes by the operating team.
  This refers to the actual time taken to complete the surgical aspect of the treatment, from the initial incision to the final suture or equivalent closing procedure.
Orthodontic Treatment Time | Treatment duration will be monitored continuously, with records updated at each patient visit.
  The time required from the initiation of orthodontic appliance placement to the achievement of the desired dental alignment and occlusion
Patient Satisfaction and Quality of Life | Surveys will be administered at 6 months and 1 year post-treatment to capture both short- term and long-term satisfaction and quality of life.
  This endpoint assesses the patient's subjective satisfaction with the treatment outcomes and the impact on their quality of life.
  Measurement Tools: Validated questionnaires such as the Oral Health Impact Profile (OHIP) and patient satisfaction surveys will be utilized.

CONTACTS AND LOCATIONS:
Locations (1):
- Dental Clinic "Dental-Service" - Department of Oral and Maxillofacial Surgery, 77 S. Vanzetti Street, Novosibirsk, Novosibirsk Oblast, Russia

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to the single-patient nature of the study and associated confidentiality limitations.